CLINICAL TRIAL: NCT02117843
Title: A Prospective, Multi-center, Single Armed Registry to Evaluate The Safety and Efficacy of 'AVI' Stent for Treating Coronary Revascularization
Brief Title: The Safety and Efficacy of 'AVI' Stent for Treating Coronary Revascularization
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Beijing AmsinoMed Medical Device Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PERFECT-I
Record Dates: First submitted 2014-04-16; First posted 2014-04-21 (Estimated); Last update posted 2017-06-27 (Actual); Status verified 2017-06

CONDITIONS: Ischemic Heart Disease; Myocardial Ischemia; Coronary Disease; Acute Coronary Syndrome
MeSH Terms: conditions — Myocardial Ischemia; Coronary Disease; Acute Coronary Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- AVI® Arsenic trioxide drug eluting stent (Experimental): The Arsenic trioxide as AVI eluting drug, biodegradable polylactic acid as drug carrier.
  Interventions: Device: AVI® Arsenic trioxide drug eluting stent

INTERVENTIONS:
Device: AVI® Arsenic trioxide drug eluting stent — AVI® Arsenic trioxide drug eluting stent

SUMMARY:
The study is a Prospective, Multi-center, Single Armed Registry to Evaluate The Safety and Efficacy of 'AVI' Stent for Treating Coronary Revascularization.

DETAILED DESCRIPTION:
The study is a Prospective, Multi-center, Single Armed Registry to Evaluate The Safety and Efficacy of 'AVI' Stent for Treating Coronary Revascularization, 1200 primary coronary artery disease patients will be enrolled, at approximately 40 sites. Subject follow-up will occur via telephone contact or clinical visit at 30 days, 6 months, 9 months, 12 months, 2-5 years after procedure.

ELIGIBILITY:
Inclusion Criteria:

Patient must be at least 18 years of age;

Ischemic heart symptom and/or myocardial ischemia, include chronic stable/unstable coronary artery disease or acute coronary syndrome(ST elevated MI and Non-ST elevated MI);

At least one lesion with a diameter stenosis >70% or more suitable for coronary stent implantation in a vessel with a reference diameter ranging from 2.5mm to 3.5mm;

If the subject has multiple vessel lesions, the implanted stents must be the same brand. The staged procedure only be allowed within 3 months after procedure, the implanted stent must be the same brand stent as the index procedure;

Subject has no CABG contraindication;

Subject or legal representative is informed the property of the study, understand the stipulations in the protocol, ensure the compliance and sign the ICF;

Exclusion Criteria:

Pregnant or nursing patients and those who plan to become pregnant up to 1 year post index procedure;

Subject has a tendency to bleeding or coagulation disorders, or has contraindication of antiplatelet and/or anticoagulant therapy, or can't accept the continue DAPT within 6 months;

Poor compliance or expectation of life less than 1 year;

Implanted any brand stent in the same target vessel within 1 year;

Left Ventricular Ejection Fraction (LVEF) of <30%;

Cardiogenic shock or haemodynamics abnormal, needs inotropic agents or mechanical support;

The subject is allergic to asprin, heparin, clopidogrel/ticlopidine, stainless steel alloy, arsenic trioxide, sirolimus, styrene-butene-styrene or polylactic acid(PLA) polymer and contrast agent;

Severe tortuous and/or heavy calcification lesion;

Two or more proximal chronic total occlusion lesion;

Bifurcation lesions with double stents;

The subject has multi-vessel lesions but can not be implanted the same brand stents;

The subject that the investigator considers he/she was unfit to implant the AVI stents and Firebird 2 stents;

The subject attended other drug/device study or in the follow-up period.

Ages: 18 Years to 76 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1200 (Estimated)
Dates: Start 2013-07; Primary Completion 2017-12 (Estimated); Study Completion 2021-04 (Estimated)

PRIMARY OUTCOMES:
Ischemia-driven target lesion failure(iTLF) , including cardiac death, target vessel related MI(Q wave and Non-Q wave) and ischemic-driven target lesion revascularization(iTLR) | at 12 months post procedure

CONTACTS AND LOCATIONS:
Overall Officials: Yitong Ma, Prof., Principal Investigator — First Affiliated Hospital of Xinjiang Medical University
Locations (1):
- The First Teaching Hospital of Xinjiang Medical University, Ürümqi, Xinjiang, China

IPD SHARING:
Plan to Share IPD: No